CLINICAL TRIAL: NCT05113394
Title: Preventing Childhood Asthma Using Prophylactic House Dust Mite Allergen Immunotherapy
Acronym: PAPA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Awaiting funding
Sponsor: Boston Children's Hospital (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other); University of North Carolina, Chapel Hill (Other); George Washington University (Other); Emory University (Other); University of Southampton (Other); Imperial College London (Other)
Responsible Party: Principal Investigator, Wanda Phipatanakul, Professor of Pediatrics, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Record Dates: First submitted 2021-10-19; First posted 2021-11-09 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Asthma; Allergy
MeSH Terms: conditions — Asthma; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Randomized (1:1), double blinded, placebo controlled, parallel arms, multi-site, Phase II study; 3 year treatment phase with further 1.5 year follow-up phase.
Who Masked: Outcomes Assessor
Masking Description: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): HDM sublingual Immunotherapy (HDM-SLIT) with Odactra® for 3 years to high-risk infants aged between 6 to 12 months at enrollment in preventing the development of asthma, assessed 1.5 years after discontinuation of treatment.
  Interventions: Drug: HDM sublingual Immunotherapy
- Placebo arm (Placebo Comparator): Placebo administered sublingually for 3 years to high-risk infants aged between 6 to 12 months with outcome of asthma development assessed 1.5 years after discontinuation of treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HDM sublingual Immunotherapy — HDM-SLIT tablet (Odactra®/Acarizax®) is a rapidly dissolving, freeze-dried, oral lyophilizate for oromucosal treatment, which contains a 1:1 mixture of two allergen extracts derived for the cultivated house dust mites, D. pteronyssinus and D. farinae. These species are included in SLIT tablet and subcutaneous immunotherapy administered for the treatment of allergic rhinitis and asthma in the pediatric and adult populations. The tablet dissolves within seconds after contact with a wet surface such as the oral mucosa. Participants will be administered the drug sublingually for 3 years.
  Other Names: dust mite sublingual immunotherapy
  Arms: Experimental arm
Drug: Placebo — Placebo sublingual therapy
  Other Names: placebo dust mite sublingual immunotherapy
  Arms: Placebo arm

SUMMARY:
To establish efficacy and safety of HDM sublingual Immunotherapy (HDM-SLIT) by comparing Odactra and placebo, when given sublingually for 3 years to high risk infants aged between 6 to 12 months at enrollment in preventing the development of asthma, assessed 1.5 years after discontinuation of treatment.

DETAILED DESCRIPTION:
Aim to prevent the development of asthma in children by intervening at a time when the developing system in still amenable to immune modulation, by using the only therapy that has proven ability to change the natural history of allergic diseases and induce clinical remission. We hypothesize that three years of HDM Immunotherapy in high-risk infants will prevent the development of asthma assessed over a period of 1.5 years after discontinuation of treatment and HDM immunotherapy will result in (a) a significant reduction in the number and pathogenic features of HDM-reactive TH2 cells, and (b) an increase in the numbers of HDM-reactive TH and TREG cells expressing the interferon-response signature. The study is a Randomized (1:1), double blinded, placebo controlled, parallel arms, multi-site, Phase II study with a 3 year treatment phase and further 1.5 year follow-up phase. The study duration for each participant is 4.5 years. Overall study duration is 84 months (7 years); which include 9 months preparation and regulatory approvals, 15 months accrual, 36 months treatment and 18 months follow-up observation period.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 6 to 12 months of age
2. history of physician diagnosed atopic dermatitis OR
3. allergen sensitization OR
4. family history of asthma or allergy

Exclusion Criteria:

1. Evidence of sensitization to house dust mite (SPT ≥3 mm OR sIgE (> 0.35 kU/L)
2. Prematurity (<37 weeks)
3. Failure to thrive
4. Need for oxygen for more than 5 days in the neonatal period
5. history of intubation or mechanical ventilation

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2027-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Asthma | 1.5 years after discontinuation of 3 years of treatment
  asthma diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Wanda Phipatanakul, MD, MS, Principal Investigator — Boston Children's Hospital